CLINICAL TRIAL: NCT01468428
Title: Small Intestinal Function in Patients With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: UAarhus - VCF
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Cystic Fibrosis; Gastrointestinal Motility
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In patients with Cystic fibrosis (CF) epithelial transport of chloride and sodium is disrupted in several organs such as airways, sweat glands, pancreas and intestines. Gastrointestinal symptoms are frequent but little is known about intestinal motility and function. Earlier studies using lactulose/hydrogen breath tests have found altered intestinal transit time. The method has several sources of errors and results have been questioned. This study is using a new, non invasive method to study intestinal motility patterns and transit times, Magnetic Tracking System - 1 (MTS-1).

The aim is to compare patterns of contractility and transit times in the stomach and small intestine in adult CF- patients with healthy controls.

Methods MTS-1 is performed without radiation and is associated with minimal discomfort for subjects. A small magnetic pill is ingest and detected by a matrix of sensors. Position and orientation of the magnet are defined by five coordinates (position: x, y, z, angle: φ, θ). Frequencies of slow waves as well as number and power of phase III contractions can be identified.

Colorectal transit times are determined with a plain abdominal x-ray. The subjects are asked to ingest a capsule containing 10 radiopaque markers on six consecutive days up to examination. The total number of markers in the entire colorectum is counted. Total transit time, as well as segmental is calculated.

Subjects 15 adult patients (> 18 years) with CF, homozygote for the mutation ΔF508, are studied. They are all pancreas insufficient (fecal elastase < 100 µg/g), with no previous intestinal resection or lung transplantation. None of them have diabetes. Patients are all in well-regulated pancreatic enzyme replacement therapy (PERT), thriving and with stabile weight over the last half year. They have had no treatment with antibiotics in the last 14 days up to the examination.

The hypothesis is that patterns of contractility and transit times are the same for CF-patients in well -regulated PERT as for healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis, severe mutations
* Pancreatic insufficiency(Fecal elastase < 100 µg/g)
* Thriving, stabile weight over the last half year
* No treatment with antibiotics in the last 14 days up to the examination

Exclusion Criteria:

* intestinal resection
* lung transplantation
* diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 15 CF patients with severe mutations and pancreatic insufficiency, without having diabetes or intestinal resection, with stable weight and no antibiotic treatment 14 days up to examination.
  * 15 age- and gender matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Small intestinal transit time
  MTS-1: A small magnet pill is ingested and its movements are monitored and recorded from mouth to caecum. The transit time of the stomach and small intestine is determined by real-time recordings.

SECONDARY OUTCOMES:
Colorectal transit time
  Colorectal transit times are obtained using a plain abdominal x-ray after subjects has ingested 10 radiopaque markers on six consecutive days up to examination. The total number of markers in the entire colorectrum is counted and total as well as segmental transit times are calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Healthy Sciencies, Aarhus, Denmark